CLINICAL TRIAL: NCT07277595
Title: KTMP: A Novel Method of Non-invasive Brain Stimulation to Enhance Motor Function in Chronic Stroke Patients.
Brief Title: kTMP in Chronic Stroke
Acronym: KULMINATE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 25-43524; R44NS139730 (NIH)
Record Dates: First submitted 2025-12-02; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Stroke; Chronic Stroke Patients; Arm Weakness as a Consequence of Stroke
Keywords: transcranial magnetic stimulation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active Treatment (Active Comparator): Active treatment with kTMP for 18 weeks
  Interventions: Device: kTMP 18 weeks
- Crossover Treatment (Other): Initial 9 weeks will receive sham kTMP treatment, followed by 9 weeks of active kTMP treatment.
  Interventions: Device: kTMP sham stimulation 9 weeks + active stimulation 9 weeks

INTERVENTIONS:
Device: kTMP sham stimulation 9 weeks + active stimulation 9 weeks — kTMP 9 weeks sham-kTMP stimulation, followed by 9 weeks active kTMP stimulation
  Arms: Crossover Treatment
Device: kTMP 18 weeks — Participants receive kTMP active stimulation for 18 weeks
  Arms: Active Treatment

SUMMARY:
kTMP, kilohertz transcutaneous magnetic perturbations, is a low intensity transcranial magnetic stimulation technique that will be used in this study to promote arm/hand rehabilitation in patients who have been disabled by stroke.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18-80 years old who have had a stroke resulting in hemiplegia
* Ability to communicate, understand, and give appropriate consent
* Other criteria may apply

Exclusion Criteria:

* Significant cognitive impairment
* inability to adhere to the study protocol or provide informed consent
* pregnancy
* additional criteria may apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2030-08-01 (Estimated); Study Completion 2030-08-01 (Estimated)

PRIMARY OUTCOMES:
Fugl Meyer Assessment | Enrollment, then weeks 3, 6, 9, 12, 15, 18, and 34.
  The Fugl-Meyer Assessment (FMA) is a structured evaluation used to measure motor recovery after a stroke, with a total score range of 0-226. Higher scores indicate better motor function, while lower scores reflect greater impairment.

SECONDARY OUTCOMES:
Wolf Motor Function Test | At enrollment, then weeks 3, 6, 9, 12, 15, 18, and 34
  Measures timed functional tasks, strength testing, and analysis of movement quality when completing various upper extremity tasks. Uses a 6 point ordinal scale (0-5), where ) is does not attempt with the involved arm and 5 is arm does participate and movement appears normal. Maximum score of 75. Lower scores indicate lower functional levels.
Stroke Impact Scale | At enrollment, then weeks 3, 6, 9, 12, 15, 18, and 34
  Self reported questionnaire that evaluates disability and health related quality of life after stroke, consisting of 59 items, assessing strength, hand function, ADL/iADL, mobility, communication, emotion, memory and thinking, participation/role function. Each item is rated in a 5 point Likert scale, where 1 equals could not do it at all and 5 equals not difficult at all. Score ranges 0-100. Higher score indicates less disability and high quality of life after stroke.
Stroke Specific QOL | At enrollment, then weeks 3, 6, 9, 12, 15, 18, and 34
  Questionnaire consisting of 49 items in the 12 domains of mobility, energy, upper extremity function, work and productivity, mood, self-care, social roles, family roles, vision, language, thinking and personality. Each item is assessed on a 5 point Guttman type scale, where 1=total help; couldn't do it at all; strongly agree and 5 =no help needed; no trouble at all; strongly disagree. Higher scores indicate better functioning.
EuroQOL | At enrollment, then weeks 3, 6, 9, 12, 15, 18, and 34
  A health questionnaire that measures 5 dimensions including mobility, self-care, usual activities, pain/discomfort, anxiety/depression. Each item is described by 3 levels of problems, where 1=none, 2=mild to moderate, and 3=severe. This provides a simple single index value for health status, where a higher score indicates worse health state.
Motor Activity Log | At enrollment, then weeks 3, 6, 9, 12, 15, 18, and 34
  Self reported perception of Quality of movement are rated in 30 functional tasks, scored on a 6 point ordinal scale where 0=weaker arm not used at all for that activity and 5=ability to use the weaker arm for that activity is as good as before the stroke(normal). A higher score indicates better quality upper extremity movement.
Modified Ashworth Scale Scores | At enrollment, then weeks 3, 6, 9, 12, 15, 18, and 34
  Test of resistance to passive movement about a joint, scores range from 0 to 5 where 0=no increase in muscle tone and 5=affected part(s) rigid. Hight scores indicate greater muscle tone.
Action Research Arm Test | At enrollment, then weeks 3, 6, 9, 12, 15, 18, and 34
  Measures performance of the upper extremity in grasp, grip, pinch, and gross arm movements, rated on a 4 point ordinal scale where 3=performs test normally and 0=can perform no part of test. Higher score indicates greater function of the upper extremity.

CONTACTS AND LOCATIONS:
Overall Officials: Karunesh Ganguly, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No